CLINICAL TRIAL: NCT00552292
Title: National Investigation of Cardiovascular Complications in Arterial Hypertension and Obesity
Brief Title: Complications in Hypertension and Obesity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Principal Investigator, Conrady Alexandra, professor, Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health
Other Study IDs: 25/1
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Metabolic Syndrome; Hypertension; Obesity; Dyslipidemia; Hyperglycemia
Keywords: metabolic syndrome; hypertension; obesity; dyslipidemia; hyperglycemia; cardiovascular complications
MeSH Terms: conditions — Metabolic Syndrome; Hypertension; Obesity; Dyslipidemias; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The study in aimed to investigate epidemiology of risk factors in Russian Federation its prognostic value aimed on acceptance of national specific definition of metabolic syndrome and guidelines for its management.

ELIGIBILITY:
Inclusion Criteria:

* Age older 18 years
* Signed informed consent
* Blood pressure more than 130 and/or 85 mm Hg
* Waist circumference more than 80 sm in females and 94 in males and/or BMI more than 25 kg/m2
* Dyslipidemia (elevated TG and/or decreased level of HDLP or therapy for high triglyceride level)
* Fasting glucose more than 5,6 mmol/l

Exclusion Criteria:

* Associated clinical conditions (stroke, TIA, MI, heart failure, renal disease, diabetes mellitus)
* Severe concomitant diseases affecting outcome

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age and sex-matched sample of subjects older 18 age
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2007-12; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
cardiovascular complications | 2007-2017

SECONDARY OUTCOMES:
diabetes mellitus | 2007-2017

CONTACTS AND LOCATIONS:
Overall Officials: Eugene V Shlyakhto, Study Director — Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health
Locations (1):
- Almazov Federal Center of Heart, Blood and Endocrinology, Saint Petersburg, Russia